CLINICAL TRIAL: NCT02719288
Title: A Multi-center, Open Label, Economic Outcome Study Comparing the Recovery of Patients Receiving CLARIX® CORD 1K as an add-on Treatment During Surgical Tendon Repair to Control Patients Receiving Standard of Care Procedures
Brief Title: Peroneal and Achilles Tendon Repair Indications With CLARIX® CORD 1K
Acronym: PATRICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amniox Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-2010
Record Dates: First submitted 2016-03-17; First posted 2016-03-25 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Peroneal and Achilles Tendon Tears

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLARIX® CORD 1K (Experimental): Applied in addition to standard of care tendon repair surgery.
  Interventions: Other: CLARIX® CORD 1K graft
- Standard of care tendon repair surgery only (No Intervention)

INTERVENTIONS:
Other: CLARIX® CORD 1K graft
  Arms: CLARIX® CORD 1K

SUMMARY:
Peroneal and Achilles tendon tears are common diseases that present challenges to surgeons due to tendon adhesion complications. Functional recovery is compromised by limiting post-operative range of motion, mobility, and can lead to considerable amount of post-operative pain for the patient.

Amniotic membrane tissue has demonstrated clinical success as an anti-inflammatory and anti-scarring agent and promoting wound healing towards regeneration.

Cryopreserved human amniotic membrane and umbilical cord (AM/UC) tissue in the form of CLARIX® CORD 1K has been used to treat over 5000 orthopedic patients. The investigators hypothesize that its use in peroneal and Achilles tendon surgical repair will enhance the overall functional recovery of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years to 80 years of age
2. Confirmed tendon pathology via MRI, if clinically necessary, with planned surgical repair that have failed conservative management (PT) for a minimum of 2 months for chronic and partial thickness tears; acute full thickness tears or tendon rupture immediately eligible.
3. Willing to follow the instructions and complete the visits required.

Exclusion Criteria:

1. Psychologically unstable
2. Acute infections that, in the opinion of the investigator, may complicate healing
3. Currently receiving chemotherapy
4. Systemic inflammatory arthritis or Rheumatoid arthritis
5. Uncontrolled diabetes as measured by A1C>12
6. Bleeding disorders
7. Unable to provide informed consent
8. Has received oral or parenteral corticosteroids or cytotoxic agents for seven consecutive days in the period of 30 days before surgery OR has received a local steroid injection within 7 days of surgery
9. Immunocompromised patients
10. Active malignancy other than non-melanoma skin cancer
11. Untreated alcohol or substance abuse issues at the time of screening
12. Pregnant women at the time of randomization
13. Currently enrolled or participated in another investigational device, drug, or biological trial within 60 days of screening
14. Allergy to amphotericin-B or Dulbecco's Modified Eagle Medium (DMEM).
15. Will undergo significant concurrent procedures with the tendon procedures on the affected foot that, in the opinion of the Investigator, may complicate healing or alter the post-operative visit schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient questionnaire describing function limitation (American Orthopaedic Foot and Ankle Society ankle hindfoot score). | Baseline and 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Scheffer Tseng, MD, PhD, Study Chair — BioTissue Holdings, Inc
Locations (4):
- United States (4):
  - Banner Estrella Medical Center, Phoenix, Arizona
  - Banner Del Webb Medical Center, Sun City West, Arizona
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Orthopedic Foot and Ankle Center, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelberman RH, Manske PR. Factors influencing flexor tendon adhesions. Hand Clin. 1985 Feb;1(1):35-42. PMID 4093463
- [Background] Adzick NS, Lorenz HP. Cells, matrix, growth factors, and the surgeon. The biology of scarless fetal wound repair. Ann Surg. 1994 Jul;220(1):10-8. doi: 10.1097/00000658-199407000-00003. PMID 8024353
- [Background] Jaibaji M. Advances in the biology of zone II flexor tendon healing and adhesion formation. Ann Plast Surg. 2000 Jul;45(1):83-92. doi: 10.1097/00000637-200045010-00017. PMID 10917106
- [Background] Liu J, Sheha H, Fu Y, Liang L, Tseng SC. Update on amniotic membrane transplantation. Expert Rev Ophthalmol. 2010 Oct;5(5):645-661. doi: 10.1586/eop.10.63. PMID 21436959
- [Background] Swift H. Amnion for leg ulcers. Lancet. 1980 Jun 21;1(8182):1366-7. doi: 10.1016/s0140-6736(80)91819-x. No abstract available. PMID 6104165
- [Background] Dua HS, Gomes JA, King AJ, Maharajan VS. The amniotic membrane in ophthalmology. Surv Ophthalmol. 2004 Jan-Feb;49(1):51-77. doi: 10.1016/j.survophthal.2003.10.004. PMID 14711440
- [Background] Bouchard CS, John T. Amniotic membrane transplantation in the management of severe ocular surface disease: indications and outcomes. Ocul Surf. 2004 Jul;2(3):201-11. doi: 10.1016/s1542-0124(12)70062-9. PMID 17216092